CLINICAL TRIAL: NCT05523219
Title: Prospective Observational Study for the Evaluation of VEOFIX Varisation Staples
Status: Completed | Type: Observational
Sponsor: Societe dEtude, de Recherche et de Fabrication (Industry)
Responsible Party: Sponsor
Other Study IDs: Veofix varisation staples
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2023-11

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This clinical investigation was led as a post-market clinical follow-up study (post-market device development stage). Therefore, its objectives were as follows:

* To assess functional clinical score's evolution,
* To evaluate patient's satisfaction
* To confirm safety of varisation staples The target population for this study was any adult patient implanted with VEOFIX varisation staples in their intended uses between 15/02/2021 and 15/05/2021.

Patients were implanted and followed as per standard of care led in the investigational site.

The following regulation and guidelines were followed for this investigation:

* Standard ISO 14155:2020 "Good Clinical Practice"undirectly applicable;
* Regulation (UE) 2016/679 (RGPD) ;
* Regulation (UE) 2017/745 (MDR) ;
* MEDDEV 2.12.1;
* Local regulation (loi " jardé ", loi " informatique et libertés "). As per its design, the investigation is considered as involving human beings, and therefore require submission to an ethic committee or declaration to a Competent Authority (ANSM) and CPP. This study was registered on CPP (CPP Ile de France VII).

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* Major patient on the date of surgery
* Patient with foot pathology requiring Akin osteotomy
* Patient not opposed to the collection of data

Exclusion Criteria:

* Patient unable to understand and follow the postoperative instructions
* Patient with a contraindication to the use of the implant
* Non-implanted patient with a varisation staple

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Due to its non-comparative design, no patient was randomized. Every patient who respected the selection criteria were included to create an exhaustive and consecutive cohort
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Victor Hugo Clinical, Paris, Île-de-France Region, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients implanted with VEOFIX varisation staples between 15/02/2021 and 15/05/2021 in Clinique Victor Hugo.
Pre-assignment Details: No SERF assembly
Groups:
- Total Cohort: The description will be carried out on the whole population really included
Period: Overall Study
Arm/Group | Total Cohort
Started | 81 (One patient was wrongly included because he did not have a SERF implant)
Completed | 73
Not Completed | 8
Not completed — Wrong inclusion | 1
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | Total Cohort
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  French nationality | 80
Side : Right, Left [Count of Participants; unit: Participants]
  Right | 51
  Left | 29
Indication : Hallux Valgus [Count of Participants; unit: Participants] | 80

OUTCOME MEASURES:

1. Primary Outcome: AOFAS Score
Description: To confirm the performance of varisation staples in conservative surgery of Hallux Valgus, according to the indications covered by the CE Marking (Akin's osteotomy) and according to the surgeon's current practice investigator.
  The scores range from 0 to 100, The average preoperative score was 50 to 60 points. Post-operatively, a score of 80 points is a good post-operative result, with the patient experiencing no or low levels of residual pain and full or partial recovery of joint function. The AOFAS Score is considered excellent between 90 and 100 points, good between 80 and 89, fair between 60 and 79, and poor below 60 points.
Time Frame: 3 and 12 months
Population: The number of scores is different for each follow-up. In fact, this score is recovered during patient follow-up.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Total Cohort
Number analyzed (Participants) | 80
points
  Preoperatively | 41.2 (17.5)
  3 months: number analyzed (Participants) | 78
  3 months | 77.0 (9.1)
  12 months: number analyzed (Participants) | 73
  12 months | 88.1 (9.4)

2. Secondary Outcome: Patient Satisfaction
Description: The information will be collected from both the patient through questionnaires to compare preoperatively situtation to last follow-up situtation
Time Frame: 3 and 12 months
Population: * 80 patients preoperatively;
  * 78 patients were available at 3 months follow-up.
  * 73 patients were available at 12 months follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Cohort
Number analyzed (Participants) | 80
Participants
  3 months: number analyzed (Participants) | 78
  3 months: Very satisfied | 17
  3 months: Satisfied | 56
  3 months: Dissatisfied | 5
  3 months: Dissappointed | 0
  12 months: number analyzed (Participants) | 73
  12 months: Very satisfied | 43
  12 months: Satisfied | 28
  12 months: Dissatisfied | 1
  12 months: Dissappointed | 1

3. Secondary Outcome: Number of Complications Observed During the Clinical Investigation
Description: Number of complications observed throughout the clinical investigation
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | Total Cohort
Number analyzed (Participants) | 80
events
  Neurogenic pain after loco-regional anaesthesia | 4
  Paraesthesia O1 | 1
  Hallux varus | 2

ADVERSE EVENTS:
Time Frame: 14.9 months
Arm/Group | Total Cohort
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 7/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Cohort (N=80)
Neurogenic pain after locoregional anaesthesia (Nervous system disorders) | 4 (4)
Paresthesia O1 (Surgical and medical procedures) | 1 (1)
Hallux Varus (Surgical and medical procedures) | 2 (2)

LIMITATIONS AND CAVEATS:
The 12 months follow-up was done in consultation, but when the patient could not move, it was done by telephone.

There is a delay in follow-ups for 12 months due to school holidays.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/19/NCT05523219/Prot_000.pdf